CLINICAL TRIAL: NCT00444860
Title: A Phase III Clinical Trial to Study the Safety, Tolerability, and Immunogenicity of ZOSTAVAX(R) in Healthy Adults in Taiwan
Brief Title: ZOSTAVAX(R) Local Registration Trial (V211-019)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V211-019; MKV211-019; 2007_008
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Varicella Virus Infection
MeSH Terms: interventions — Herpes Zoster Vaccine

ARMS (1):
- 1 (Experimental): Zostavax
  Interventions: Biological: Zoster Vaccine, Live, (Oka-Merck)

INTERVENTIONS:
Biological: Zoster Vaccine, Live, (Oka-Merck) — A single dose of 0.65 ml of Zostavax injection was given to each study subject
  Other Names: Zostavax

SUMMARY:
The purpose of this study is to obtain safety and immunogenicity data for the refrigerator-stable formulation of ZOSTAVAX(R) in taiwanese adults.

ELIGIBILITY:
Inclusion Criteria:

* Subject Is Older Than 50 Years Of Age On Day Of Signing Informed Consent
* All Females Must Be Postmenopausal Or Have A Negative Serum Or Urine Pregnancy Test

  * Postmenopausal Is Defined As 6 Months Of Spontaneous Amenorrhea With Serum Follicle Stimulating Hormone (Fsh) Levels In The Postmenopausal Range As Determined By The Laboratory, Or 12 Months Of Spontaneous Amenorrhea
* A Subject Who Is Of Reproductive Potential Must Agree To Remain Abstinent Or Use (Or Have Her Partner Use) 2 Acceptable Methods Of Birth Control For Three Months After Vaccination

  * Acceptable Methods Of Birth Control Are: Intrauterine Device, Diaphragm With Spermicide, Contraceptive Sponge, Oral Contraceptive Pills, Condom, Tubal Ligation, And Vasectomy
* Subject Must Sign Informed Consent Prior To Any Study Procedure
* Subject Must Be afebrile (<38.3 °C Oral) On Day Of Vaccination
* Any Underlying Chronic Illness Must Be In Stable Condition

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-03; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The geometric mean fold rise (GMFR) of subjects VZV antibody titers from prevaccination to 4 weeks postvaccination, and the geometric mean titers (GMTs) at prevaccination and 4 weeks postvaccination, as measured by gpELISA, will be assessed. | prevaccination and 4 weeks postvaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Yao CA, Chen LK, Huang KC. The immunogenicity and safety of zoster vaccine in Taiwanese adults. Vaccine. 2015 Mar 24;33(13):1515-7. doi: 10.1016/j.vaccine.2015.01.085. Epub 2015 Feb 11. PMID 25681662